CLINICAL TRIAL: NCT06894875
Title: Examining the Safety and Tolerability of Lentil Protein Hydrolysate in Healthy Males and Females Whilst Exploring the Effects of a Dose Range on Blood Pressure Control and Vascular Function and Exercise Performance
Brief Title: Effects of Lentil Protein Hydrolysate on Blood Pressure Control, Vascular Function and Exercise Performance
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Nuritas Ltd (Industry)
Collaborators: Australian Catholic University (Other); Baker Heart and Diabetes Institute (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Other
Other Study IDs: PEPLEN24
Record Dates: First submitted 2025-03-10; First posted 2025-03-25 (Actual); Last update posted 2025-12-16 (Actual); Status verified 2025-12

CONDITIONS: Exercise; Blood Pressure; Vasodilation; Vascular Function in Healthy Volunteers; Exercise Performance; Safety and Tolerability in Healthy Volunteers
Keywords: Exercise performance; Vascular function; blood pressure control; Lentil protein hydrolysate
MeSH Terms: conditions — Motor Activity; Aneurysm

STUDY DESIGN:
Intervention Model Description: Randomized, double-blind, placebo-controlled, parallel dose response study conducted over 28 days
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Lentil protein hydrolysate 500 mg/day (Experimental)
  Interventions: Dietary Supplement: Lentil protein hydrolysate
- Lentil protein hydrolysate 1000 mg/day (Experimental)
  Interventions: Dietary Supplement: Lentil protein hydrolysate
- Lentil protein hydrolysate 2000 mg/day (Experimental)
  Interventions: Dietary Supplement: Lentil protein hydrolysate
- Microcrystalline Cellulose 2000mg/day (Placebo Comparator)
  Interventions: Dietary Supplement: Placebo MCC micro-crystalline cellulose

INTERVENTIONS:
Dietary Supplement: Lentil protein hydrolysate — Plant protein hydrolysate
  Arms: Lentil protein hydrolysate 1000 mg/day; Lentil protein hydrolysate 2000 mg/day; Lentil protein hydrolysate 500 mg/day
Dietary Supplement: Placebo MCC micro-crystalline cellulose — Placebo MCC micro-crystalline cellulose
  Arms: Microcrystalline Cellulose 2000mg/day

SUMMARY:
Examining the safety and tolerability of Lentil Protein Hydrolysate in healthy males and females whilst exploring the effects of a dose range on blood pressure control and vascular function and exercise performance

DETAILED DESCRIPTION:
The aim of this trial is to evaluate the safety and tolerability of a lentil protein hydrolysate (LPH) in healthy participants while exploring effects on blood pressure control, vascular function and exercise performance. The study will be conducted in men and women over 4 weeks.

Specifically, the study has three key objectives:

1. To determine the safety and tolerability of 500 - 2000mg of a novel plant-based supplement LPH) in healthy volunteers as assessed via AE reporting, changes in clinic blood pressure and supplementation induced orthostatic hypotension during a sit-to-stand challenge.
2. To explore the effects of 4-weeks of lentil protein hydrolysate supplementation on markers of vascular age and endothelial function, fatigue, quality of life, and grip strength.
3. To explore the effects of 4-weeks of LPH supplementation on markers of exercise performance, including cardiorespiratory fitness (VO2max) and substrate utilisation during sub-maximal, steady-state exercise. This trial incorporates a wearable device to measure physical activity, cardiac health, sleep metrics and heart rate variability.

ELIGIBILITY:
Inclusion Criteria:

* Willing to provide written and dated informed consent to participate in the study.
* Willing and able to comply with the protocol.
* Are not on any medication, or supplements which would impact the trial in the opinions of the investigator or Sponsor.
* Male or female between 18 and 45 years of age (18.5 kg/m2 ≥ BMI < 30 kg/m2).
* Comply with ACSM guidelines for physical activity.
* Have not participated in a clinical trial within the past month and agree to not participate in another clinical trial during the study period.
* Agree to not significantly alter diet or exercise routine during the trial period.
* Willing to wear a wearable device continuously for the duration of the study

Exclusion Criteria:

* Subjects having a known allergy or hypersensitivity to any of the ingredients in the investigational products.
* Subjects with a history of alcohol and/or other drug abuse in the past year.
* Has performed strenuous exercise (rating of perceived exertion ≥ 13) ≤ 48 hours before laboratory visit (Borg, 1982).
* Consuming >14 alcoholic drinks per week or > 2 drinks/day in the 48 hours preceding a clinic visit.
* Active smokers, nicotine use or vaping
* Subjects suffering from a sleep disorder and/or who have a known history of (or was being treated for) clinical depression, eating disorder(s) or any other psychiatric condition(s) that might put the subject at risk and/or confounded the results of the study.
* Subjects with a history of being diagnosed with phenylketonuria or another disease affecting amino acid metabolism (i.e., maple syrup urine disease, etc.).
* Subjects with an elevated resting heart rate (>100 bpm) or blood pressure (systolic BP >140 mmHg or diastolic BP >90 mmHg).
* Pregnant or lactating women
* Presentation of orthostatic hypotension during the screening and familiarisation study visit
* Any condition which in the opinion of the investigator makes the participant unsuitable for inclusion.

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 48 (Estimated)
Dates: Start 2025-06-24 (Actual); Primary Completion 2025-12-24 (Estimated); Study Completion 2026-03-30 (Estimated)

PRIMARY OUTCOMES:
Safety and Tolerability of a dose range of Lentil protein hydrolyste via adverse event reporting | Day 1 to Day 28
  Change from baseline to the end of the study period in safety via adverse event frequency and severity between placebo and a dose range of Lentil protein hydrolysate

SECONDARY OUTCOMES:
Safety and Tolerability of a dose range of Lentil protein hydrolyste via blood pressure recording | Day 1 to Day 28
  Elevation in resting systolic or diastolic blood pressure >10mm Hg between baseline and after supplementation with lentil protein hydrolysate or placebo.
Safety and Tolerability of a dose range of Lentil protein hydrolyste via blood pressure recording | Day 1
  Decrease in systolic (>20mmHg) or diastolic (>10mmHg) blood pressure upon standing after acute supplementation with lentil protein hydrolysate or placebo.
Safety via electrolytes and liver function tests | Day 1 to Day 28
  Change from baseline to the end of the study period in safety determined by combining results of a full blood test investigating concentration (cells/L) and quantity of red blood cells, white blood cells and platelets, electrolytes (mmol/L) and concentrations of liver function markers (U/L); Albumin, Bilirubin, Alanine aminotransferase (ALT), Aspartate amino transferase (AST), Gamma-glutamyl transferase (GGT) and Alkaline phosphatase (ALP)
Arterial stiffness | Day 1 to Day 28
  Change from baseline to the end of the study period in central arterial stiffness, measured via aortic pulse-wave velocity
Endothelial function | Day 1 to Day 28
  Change from baseline to the end of the study period in endothelium-dependent vascular function measured by flow-mediated dilation
Substrate utilisation during sub-maximal, steady-state exercise | Day 1 to Day 28
  Change from baseline to the end of the study period in the rate of oxygen consumption and the oxidative rate of fat and carbohydrates during steady-state exercise
Cardiorespiratory fitness (VO2max) | Day 1 to Day 28
  Change from baseline to the end of the study period in cardiorespiratory fitness measured during a cardiopulmonary exercise test
Blood pressure response to exercise | Day 1 to Day 28
  Change from baseline to the end of the study period in blood pressure response to cardiopulmonary exercise test
Quality of life via 12-item Short-Form Health Survey version 2 | Day 1 to Day 28
  Change from baseline to the end of the study period in general health via 12-item Short-Form Health Survey version 2
Fatigue symptoms via Multidimensional Fatigue Inventory | Day 1 to Day 28
  Change from baseline to the end of the study period in fatigue symptoms measured via Multidimensional Fatigue Inventory where scores range from 1 (no fatigue) to 50 (severe fatigue)
Grip Strength | Day 1 to Day 28
  Change from baseline to the end of the study period in hand grip strength measured via a hand-held dynamometer
Markers associated with inflammation via blood test | Day 1 to Day 28
  Change from baseline to the end of the study period in inflammatory Markers such as CRP

OTHER OUTCOMES:
Habitual physical activity via wearable device | Day 1 to Day 28
  Change from baseline to the end of the study period in habitual physical activity measured via a 3D accelerometer
Sleep biometrics via wearable device | Day 1 to Day 28
  Change from baseline to the end of the study period in biometric measures of sleep quality including heart rate (BPM), heart rate variability (RMSSD) and phases of sleep (mins in REM, deep and light) which will be combined to assess overall impact on sleep score (0-100) and readiness score (0-100).

CONTACTS AND LOCATIONS:
Locations (1):
- Baker Heart and Diabetes Institute, Melbourne, Victoria, Australia

IPD SHARING:
Plan to Share IPD: No